CLINICAL TRIAL: NCT02969213
Title: Big Data Construction and Biological Etiological Epidemiology Study of Children Epilepsy in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ling Li, chief physician,proffessor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XH-16-029
Record Dates: First submitted 2016-10-19; First posted 2016-11-21 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Epilepsy
Keywords: Electronic management of epilepsy; biological etiology; Chinese children
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Genetic: patients with Gene detection (+)
- Metabolism: patients with Metabolic disturbance
- Immune: patients with Immunological marker and Immunotherapy (+)
- infection: patients with the Infection of central nervous system
- structure: patients with abnormal image of brain
- unknown: patients not found any reason

SUMMARY:
The purpose of this study is to develop the electronic management platform for children with epilepsy, establish large data of Chinese children with epilepsy and explore its biological etiology.

DETAILED DESCRIPTION:
The establishment of the electronic management platform for children with epilepsy and large data of epilepsy in Chinese children as well as the epidemiological study its biological etiology.

ELIGIBILITY:
Inclusion Criteria:

* Children with epilepsy diagnosis, seizure types and causes of disease classification in accordance with the International Association for the diagnosis and treatment of epilepsy in 2015 guidelines
* Epilepsy children Included 0-14 years old from outpatients and inpatients by the Children's epilepsy specialist using iGrowSys management platform and clinical research, and medical records data entry complete in all China

Exclusion Criteria:

* The patients that recorded data is not complete, telephone and communication address unknown
* The patients that families do not have Internet or children and families will not access the Internet, can not be online operation

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 0-14 years old epilepsy patients in China
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The data of over 10 thousand childhood epilepsy patients in China | 26 month after developing a public platform for electronic analysis and management
  To develop a public platform for electronic analysis and management of children epilepsy to doctors and patients in China

SECONDARY OUTCOMES:
Incidence of several different causes of children epilepsy in China | up to 26 months
  A surveillance mechanism will be developed to identify and recruit children with epilepsy from the public platform for electronic analysis management of children epilepsy for doctors and patients

OTHER OUTCOMES:
gene mutation | 30 days after receipt of DNA sample
  To detect the mutation and characterize the genetic architecture and risk variants of epilepsy using genomic methods
immune factors | 7days after receipt of blood sample or/and cerebrospinal fluid
  To test Inflammatory factors, Autoimmune antibodies , Immunoglobulin
metabolic factors | 7days after receipt of blood sample or/and urine
  To test tandem mass spectrometry and enzyme
structural factors | 5ays after patients see doctor
  To scan head MRI
Infection factors | 7days after receipt of blood sample, urine and cerebrospinal fluid
  To test various pathogen

CONTACTS AND LOCATIONS:
Locations (1):
- Ling Li, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sauro KM, Wiebe S, Dunkley C, Janszky J, Kumlien E, Moshe S, Nakasato N, Pedley TA, Perucca E, Senties H, Thomas SV, Wang Y, Wilmshurst J, Jette N. The current state of epilepsy guidelines: A systematic review. Epilepsia. 2016 Jan;57(1):13-23. doi: 10.1111/epi.13273. Epub 2015 Dec 10. PMID 26659723
- [Result] Singh A, Trevick S. The Epidemiology of Global Epilepsy. Neurol Clin. 2016 Nov;34(4):837-847. doi: 10.1016/j.ncl.2016.06.015. PMID 27719996
- [Result] Lua PL, Neni WS. Health-related quality of life improvement via telemedicine for epilepsy: printed versus SMS-based education intervention. Qual Life Res. 2013 Oct;22(8):2123-32. doi: 10.1007/s11136-013-0352-6. Epub 2013 Jan 18. PMID 23329469
- [Result] Coles LD, Patterson EE, Sheffield WD, Mavoori J, Higgins J, Michael B, Leyde K, Cloyd JC, Litt B, Vite C, Worrell GA. Feasibility study of a caregiver seizure alert system in canine epilepsy. Epilepsy Res. 2013 Oct;106(3):456-60. doi: 10.1016/j.eplepsyres.2013.06.007. Epub 2013 Aug 18. PMID 23962794
- [Result] Tzallas AT, Tsipouras MG, Rigas G, Tsalikakis DG, Karvounis EC, Chondrogiorgi M, Psomadellis F, Cancela J, Pastorino M, Waldmeyer MT, Konitsiotis S, Fotiadis DI. PERFORM: a system for monitoring, assessment and management of patients with Parkinson's disease. Sensors (Basel). 2014 Nov 11;14(11):21329-57. doi: 10.3390/s141121329. PMID 25393786
- [Result] Larner AJ. Teleneurology: an overview of current status. Pract Neurol. 2011 Oct;11(5):283-8. doi: 10.1136/practneurol-2011-000090. PMID 21921003
- [Result] Hani AJ, Mikati HM, Mikati MA. Genetics of pediatric epilepsy. Pediatr Clin North Am. 2015 Jun;62(3):703-22. doi: 10.1016/j.pcl.2015.03.013. PMID 26022171
- [Result] Bearden D, Strong A, Ehnot J, DiGiovine M, Dlugos D, Goldberg EM. Targeted treatment of migrating partial seizures of infancy with quinidine. Ann Neurol. 2014 Sep;76(3):457-61. doi: 10.1002/ana.24229. Epub 2014 Jul 26. PMID 25042079
- [Result] Wright S, Vincent A. Progress in autoimmune epileptic encephalitis. Curr Opin Neurol. 2016 Apr;29(2):151-7. doi: 10.1097/WCO.0000000000000304. PMID 26886357
- [Result] Patel J, Mercimek-Mahmutoglu S. Epileptic Encephalopathy in Childhood: A Stepwise Approach for Identification of Underlying Genetic Causes. Indian J Pediatr. 2016 Oct;83(10):1164-74. doi: 10.1007/s12098-015-1979-9. Epub 2016 Jan 29. PMID 26821542
- [Result] Kim EH, Ko TS. Cognitive impairment in childhood onset epilepsy: up-to-date information about its causes. Korean J Pediatr. 2016 Apr;59(4):155-64. doi: 10.3345/kjp.2016.59.4.155. Epub 2016 Apr 30. PMID 27186225
- [Result] Bonello M, Michael BD, Solomon T. Infective Causes of Epilepsy. Semin Neurol. 2015 Jun;35(3):235-44. doi: 10.1055/s-0035-1552619. Epub 2015 Jun 10. PMID 26060903
- [Derived] Zhang Z, Wu J, Xu D, Zhao S, Lian D, Zhang D, Li L. Clinical characteristics and immunotherapy efficacy in autoimmune-associated benign epilepsy with centrotemporal spikes: A prospective cohort study. J Neuroimmunol. 2025 Jul 15;404:578603. doi: 10.1016/j.jneuroim.2025.578603. Epub 2025 Apr 4. PMID 40209515
- [Derived] Yin Y, Wu J, Wu S, Chen S, Cheng W, Li L, Wang H. Usefulness of brain FDG PET/CT imaging in pediatric patients with suspected autoimmune encephalitis from a prospective study. Eur J Nucl Med Mol Imaging. 2022 May;49(6):1918-1929. doi: 10.1007/s00259-021-05649-w. Epub 2021 Dec 23. PMID 34939173